CLINICAL TRIAL: NCT03832842
Title: Thrombin Generation as a New Test for Anticoagulation Management in Patients With ECMO
Acronym: ECMOstase
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7251
Record Dates: First submitted 2019-01-23; First posted 2019-02-06 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Implantation of a Veno-arterial or Veno-venous ECMO
Keywords: ECMO; thrombin generation test; hemostasis; bleeding events; thrombotic events
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and serum will be sampled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample

SUMMARY:
ECMO (Extracorporeal Membrane Oxygenation) is a circulatory assistance device aiming at maintaining or restoring cardiopulmonary circulation. Complications of this device are mainly hemorrhagic, related to coagulopathy induced by the initial pathology or by the device itself, or thrombotic and ischemic. One of the major challenges is therefore the management of a suitable curative anticoagulation, sufficient to limit the activation of hemostasis du to the ECMO, but reasonable to prevent hemorrhagic complications. To date, there is no standardized and validated protocol for the management of anticoagulation of patients under ECMO. The thrombin generation may be a valuable test to manage anticoagulation of patients with ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years old
* Implantation of a veno-arterial or veno-venous ECMO during hospitalization in intensive care
* Informed consent

Exclusion Criteria:

* Patient on veno-arterial ECMO after cardiac, cardiopulmonary surgery or after insertion of a left or biventricular cardiac assist device
* Contraindication to curative anticoagulation
* Congenital hemostasis disorder or anatomical abnormality predisposing to hemorrhage (hemophilia, constitutional thrombocytopathies, Willebrand disease, hereditary hemorrhagic telangiectasia, etc.)
* History of heparin-induced thrombocytopenia
* Moribund patient at the day of inclusion
* Do Not Resuscitate decision
* Subject under the protection of justice
* Subject under guardianship or curatorship
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Implantation of a veno-arterial or veno-venous ECMO during hospitalization in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
The endogenous thrombin potential (ETP) will be measured. | prior to ECMO placement at Hours 0 (ECMO circulation)
The endogenous thrombin potential (ETP) will be measured. | Hours 12
The endogenous thrombin potential (ETP) will be measured. | daily from Day1 to Day10 and at each dosing of anti-Xa.

SECONDARY OUTCOMES:
Levels of hemostasis parameters: | daily from Day1 to Day10
  thrombin generation test
Levels of hemostasis parameters: | daily from Day1 to Day10
  platelets
Levels of hemostasis parameters: | daily from Day1 to Day10
  anti-Xa
Levels of hemostasis parameters: | daily from Day1 to Day10
  aPTT
Levels of hemostasis parameters: | daily from Day1 to Day10
  prothrombin time
Levels of hemostasis parameters: | daily from Day1 to Day10
  fibrinogen
Levels of hemostasis parameters: | daily from Day1 to Day10
  factor V
Levels of hemostasis parameters: | daily from Day1 to Day10
  D-dimers
Levels of hemostasis parameters: | daily from Day1 to Day10
  antithrombin
Levels of markers of vascular cell activation | daily from Day1 to Day10
  microvesicles
Levels of markers of vascular cell activation | daily from Day1 to Day10
  neutrophil extra-cellular traps
Incidence of bleeding events defined by the WHO classification, | daily from Day1 to Day10
  type of bleeding (venous or arterial), blood/platelet/plasma transfusion (number, volume), fibrinogen treatment, calcium treatment, therapeutic intervention (surgical/radiological/endoscopic/manual)
Incidence of thrombotic and ischemic events: ischemic stroke, limb ischemia, myocardial infarction, ECMO thrombosis | daily from Day1 to Day10
Mortality: number of patients who are dead by day 28 | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Julie HELMS, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Réanimation médicale CHU Strasbourg, Strasbourg, France